CLINICAL TRIAL: NCT01362179
Title: Incidence of Hematologic and Non-Hematologic Malignancies, Thrombotic Events, and Autoimmune Disorders in Unrelated Normal Donors Undergoing Bone Marrow Harvest Versus Peripheral Blood Stem Cell Mobilization With Recombinant Human Granulocyte Colony-Stimulating Factor (rHuG-CSF)
Brief Title: National Marrow Donor Program Long-Term Donor Follow-Up
Acronym: LTDFU
Status: Completed | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other)
Responsible Party: Sponsor
Other Study IDs: LTDFU
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-03

CONDITIONS: Hematologic Neoplasms
Keywords: malignant myeloid hematologic disorders; filgrastim; long term incidence; donors who received and in those who did not receive filgrastim.
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- unstimulated BM donors: Observational (non-interventional) study.
- filgrastim-mobilized PBSC donors: Observational (non-interventional) study.

SUMMARY:
This is an observational study of unstimulated bone marrow (BM) and filgrastim-mobilized peripheral blood stem cell (PBSC) donors. The primary goal is to evaluate the hypothesis that the incidence of targeted malignant, thrombotic and autoimmune disorders after unrelated hematopoietic stem cell donation are similar between unstimulated BM and filgrastim-mobilized PBSC donors.

DETAILED DESCRIPTION:
This is an observational study of unstimulated bone marrow (BM) and filgrastim-mobilized peripheral blood stem cell (PBSC) donors. The primary goal is to evaluate the hypothesis that the incidence of targeted malignant, thrombotic and autoimmune disorders after unrelated hematopoietic stem cell donation are similar between unstimulated BM and filgrastim-mobilized PBSC donors. Donors will undergo biennial surveys until study completion. Cases of targeted disorders will be reviewed by the medical monitors to confirm the veracity of the report.

ELIGIBILITY:
Inclusion Criteria:

1. Unrelated donor who donated either unstimulated BM or filgrastim-mobilized PBSC between July 1, 1999 and approximately five years post study activation.
2. Unrelated donor who received at least one injection of filgrastim or more, but did not donate filgrastim-mobilized PBSC between July 1, 1999 and approximately five years post study activation.
3. Donation was managed by a U.S. NMDP donor center.
4. Signed informed consent for participation in this long-term donor follow-up study. Concurrent enrollment on other studies is permitted.

Exclusion Criteria:

1. Unrelated donor who donated filgrastim-mobilized bone marrow.
2. Donation was managed by a non-U.S. donor center.
3. Donor is unable to verbally communicate in any of the following languages: English, Spanish, Mandarin Chinese, Cantonese Chinese, Vietnamese, Korean, or Portuguese.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 10,000 unstimulated BM donors and 20,000 filgrastim-mobilized PBSC donors
Sampling Method: Non-Probability Sample
Enrollment: 21974 (Actual)
Dates: Start 2010-10; Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Incidence of malignant myeloid hematologic disorders | Post HSCT donation
  To describe the long-term incidence of malignant myeloid hematologic disorders in donors who received and in those who did not receive filgrastim.

CONTACTS AND LOCATIONS:
Overall Officials: John P Miller, MD, PhD, Principal Investigator — National Marrow Donor Program
Locations (29):
- United States (28):
  - City of Hope, Duarte, California
  - National Marrow Donor Program Northern California & Northwest District, Oakland, California
  - National Marrow Donor Program Southern California & Southwest District, Santa Ana, California
  - Colorado Marrow Donor Program, Denver, Colorado
  - OneBlood, Fort Lauderdale, Florida
  - Hawaii Bone Marrow Donor Registry, Honolulu, Hawaii
  - LifeSource, Glenview, Illinois
  - Rock River Valley Blood Center, Rockford, Illinois
  - Indiana Blood Center, Indianapolis, Indiana
  - National Marrow Donor Program Southcentral District, Heart of America, Leawood, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Michigan Blood, Grand Rapids, Michigan
  - The HLA Registry, Oradell, New Jersey
  - New York Blood Center, Brooklyn, New York
  - DKMS Americas, New York, New York
  - National Marrow Donor Program Southeast District, Charlotte, North Carolina
  - National Marrow Donor Program Northcentral District, Cleveland, Ohio
  - Oklahoma Blood Institute, Oklahoma City, Oklahoma
  - National Marrow Donor Program Northeast District, Philadelphia, Pennsylvania
  - Rhode Island Blood Center, Providence, Rhode Island
  - Blood Assurance, Inc., Chattanooga, Tennessee
  - Cooperative Appalachian Marrow Program Medic Regional Blood Center, Knoxville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - Cook Children's, El Paso, Texas
  - Gulf Coast Regional Blood Center, Houston, Texas
  - South Texas Blood and Tissue Center, San Antonio, Texas
  - Scott & White Clinic, Temple, Texas
  - Community Blood Center, Inc., Appleton, Wisconsin
- National Marrow Donor Program at Puerto Rico, Guaynabo, PR, Puerto Rico